CLINICAL TRIAL: NCT05345457
Title: Outpatient Antibiotics Following Previable Rupture of Membranes (pPPROM) Between 18 0/7 and 22 6/7 Weeks Gestational Age
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: MetroHealth Medical Center (Other); The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, David Hackney MD, MS, Division Director, Maternal-Fetal Medicine, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY20220251
Record Dates: First submitted 2022-04-14; First posted 2022-04-26 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Pregnancy Preterm; Pregnancy Prom; PROM, Preterm (Pregnancy); PROM (Pregnancy); Premat Rupture Membranes Preterm Unspec to Length of Time Between Rupture/Labor; Premature Birth
MeSH Terms: conditions — Fetal Membranes, Premature Rupture; Premature Birth | interventions — Azithromycin; Amoxicillin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Antibiotics (Experimental): Patients randomized into the treatment (i.e., antibiotics) arm of the study will be treated with a seven-day course of oral azithromycin and amoxicillin. Azithromycin will be dosed as single 500 mg dose (2-250mg oral tablets) administered immediately following randomization, yet prior to discharge to home, followed with 1-250mg oral tablet daily for 4 additional days (for a total of 5 days). Amoxicillin will be dosed as a single-500mg oral tablet three times daily for 7 days with first dose also being given prior to discharge home.
  Interventions: Drug: Azithromycin Pill; Drug: Amoxicillin Pill
- No antibiotics (No Intervention): Patients randomized into the control (i.e., no antibiotics arm) will be managed according to standard of care practices for previable PPROM desiring of expectant management.

INTERVENTIONS:
Drug: Azithromycin Pill — Azithromycin will be dosed as single 500 mg dose (2-250mg oral tablets) administered immediately following randomization, yet prior to discharge to home, followed with 1-250mg oral tablet daily for 4 additional days (for a total of 5 days).
  Arms: Antibiotics
Drug: Amoxicillin Pill — Amoxicillin will be dosed as a single-500mg oral tablet three times daily for 7 days with first dose also being given prior to discharge home.
  Arms: Antibiotics

SUMMARY:
A randomized, controlled, non-placebo trial to primarily assess the effect of oral, outpatient antibiotics (i.e., azithromycin and amoxicillin) on latency (i.e., proportion of patients that deliver within 28 days from membrane rupture) following previable, prelabor rupture of membranes between 18 0/7 and 22 6/7 weeks gestational age.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* Pregnant
* Live, singleton gestation
* Patient able to provide informed consent
* Gestational age between 18 weeks and 0 days and 22 weeks and 6 days at the time of -membrane rupture
* Diagnosis of preterm, prelabor rupture of membranes by clinical exam findings of either 1) visualization of amniotic fluid passing from the cervical canal and/or pooling in the vagina via sterile speculum examination, 2) a basic pH (i.e., positive nitrazine) test of vaginal fluid, 3) arborization (i.e., ferning) of dried vaginal fluid identified via microscopic examination, and/or 4) an amniotic fluid index (AFI) of less than 4cm

Exclusion Criteria:

* Gestational dating performed or confirmed by ultrasound at ≥ 18 weeks and 0 days gestational age
* Patient desires pregnancy interruption or induction of labor
* Known major fetal anomaly or aneuploidy
* Amniocentesis ≤ 7 days of diagnosis of rupture of membranes
* Cervical cerclage placement ≤ 7 days of diagnosis of rupture of membranes
* Known drug allergy or significant adverse reactions to macrolide or penicillin antibiotics
* Current antibiotic use at the time of membrane rupture diagnosis
* Vaginal bleeding at the time of membrane rupture diagnosis or within first 24 hours from diagnosis
* Febrile at the time of membrane rupture diagnosis (i.e., temperature ≥ 38 degrees Celsius) and/or within first 24 hours of diagnosis
* Active preterm labor at the time of membrane rupture diagnosis (i.e., consistent contraction pattern associated with cervical change) and/or within first 24 hours of diagnosis
* Cervical dilation of ≥ 4 cm
* Prolapse of fetal parts beyond the level of the internal cervical os
* Declination to complete full, 7-day outpatient monitoring prior to hospital re-admission should rupture occur during the 22nd week of gestation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2023-01-13 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Delivery within 28 days | 28 days from date of rupture
  The proportion of patients that undergo a spontaneous or medically-indicated delivery within 28 days from diagnosis of previable prelabor rupture of membranes (pPPROM)

SECONDARY OUTCOMES:
Severe maternal morbidity composite | From diagnosis of membrane rupture to 6 weeks following delivery
  The proportion of patient's "positive" for severe maternal morbidity composite. A patient will be termed "positive" for severe maternal morbidity composite if any one of the following is diagnosed: maternal sepsis, postpartum hemorrhage, maternal ICU admission, maternal death.
Severe neonatal morbidity composite | From date of delivery to date of hospital discharge (up to 6 months)
  The proportion of patient's "positive" for severe neonatal morbidity composite. A neonate will be termed "positive" for severe neonatal morbidity composite if any one of the following is diagnosis: bronchopulmonary dysplasia (BPD), pulmonary hypoplasia, intraventricular hemorrhage (IVH) grade III/IV, necrotizing enterocolitis (NEC) Bell's Stage II or greater, neonatal sepsis with positive blood cultures, neonatal pneumonia with positive blood cultures, neonatal death.

CONTACTS AND LOCATIONS:
Overall Officials: David Hackney, MD, Principal Investigator — University Hospitals Cleveland Medical Center; Justin Lappen, MD, Principal Investigator — The Cleveland Clinic; Brian Mercer, MD, Principal Investigator — MetroHealth Hospitals
Locations (3):
- United States (3):
  - University Hospitals, Cleveland, Ohio
  - MetroHealth, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: Yes
Once data collection and primary analysis has been completed. A de-identified data set will be provided.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will become available upon publication of study results and remain available for 2 years upon study completion.

REFERENCES:
- [Background] Martin JA, Hamilton BE, Ventura SJ, Osterman MJ, Wilson EC, Mathews TJ. Births: final data for 2010. Natl Vital Stat Rep. 2012 Aug 28;61(1):1-72. PMID 24974589
- [Background] Mathews TJ, MacDorman MF. Infant mortality statistics from the 2006 period linked birth/infant death data set. Natl Vital Stat Rep. 2010 Apr 30;58(17):1-31. PMID 20815136
- [Background] Waters TP, Mercer B. Preterm PROM: prediction, prevention, principles. Clin Obstet Gynecol. 2011 Jun;54(2):307-12. doi: 10.1097/GRF.0b013e318217d4d3. PMID 21508700
- [Background] Kilbride HW, Thibeault DW. Neonatal complications of preterm premature rupture of membranes. Pathophysiology and management. Clin Perinatol. 2001 Dec;28(4):761-85. doi: 10.1016/s0095-5108(03)00076-9. PMID 11817188
- [Background] Yeast JD. Preterm premature rupture of the membranes before viability. Clin Perinatol. 2001 Dec;28(4):849-60. doi: 10.1016/s0095-5108(03)00082-4. PMID 11758532
- [Background] Muris C, Girard B, Creveuil C, Durin L, Herlicoviez M, Dreyfus M. Management of premature rupture of membranes before 25 weeks. Eur J Obstet Gynecol Reprod Biol. 2007 Apr;131(2):163-8. doi: 10.1016/j.ejogrb.2006.05.016. Epub 2006 Jul 17. PMID 16846673
- [Background] Mercer BM, Miodovnik M, Thurnau GR, Goldenberg RL, Das AF, Ramsey RD, Rabello YA, Meis PJ, Moawad AH, Iams JD, Van Dorsten JP, Paul RH, Bottoms SF, Merenstein G, Thom EA, Roberts JM, McNellis D. Antibiotic therapy for reduction of infant morbidity after preterm premature rupture of the membranes. A randomized controlled trial. National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. JAMA. 1997 Sep 24;278(12):989-95. PMID 9307346
- [Background] American College of Obstetricians and Gynecologists; Society for Maternal-Fetal Medicine. Obstetric Care consensus No. 6: Periviable Birth. Obstet Gynecol. 2017 Oct;130(4):e187-e199. doi: 10.1097/AOG.0000000000002352. PMID 28937572
- [Background] Grisaru-Granovsky S, Eitan R, Kaplan M, Samueloff A. Expectant management of midtrimester premature rupture of membranes: a plea for limits. J Perinatol. 2003 Apr-May;23(3):235-9. doi: 10.1038/sj.jp.7210880. PMID 12732862
- [Background] Schucker JL, Mercer BM. Midtrimester premature rupture of the membranes. Semin Perinatol. 1996 Oct;20(5):389-400. doi: 10.1016/s0146-0005(96)80006-1. PMID 8912993
- [Background] Waters TP, Mercer BM. The management of preterm premature rupture of the membranes near the limit of fetal viability. Am J Obstet Gynecol. 2009 Sep;201(3):230-40. doi: 10.1016/j.ajog.2009.06.049. PMID 19733274
- [Background] Pristauz G, Bauer M, Maurer-Fellbaum U, Rotky-Fast C, Bader AA, Haas J, Lang U. Neonatal outcome and two-year follow-up after expectant management of second trimester rupture of membranes. Int J Gynaecol Obstet. 2008 Jun;101(3):264-8. doi: 10.1016/j.ijgo.2007.12.007. Epub 2008 Mar 4. PMID 18289539
- [Background] Dotters-Katz SK, Myrick O, Smid M, Manuck TA, Boggess KA, Goodnight W. Use of prophylactic antibiotics in women with previable prelabor rupture of membranes. J Neonatal Perinatal Med. 2017;10(4):431-437. doi: 10.3233/NPM-16165. PMID 29286934
- [Background] Manuck TA, Eller AG, Esplin MS, Stoddard GJ, Varner MW, Silver RM. Outcomes of expectantly managed preterm premature rupture of membranes occurring before 24 weeks of gestation. Obstet Gynecol. 2009 Jul;114(1):29-37. doi: 10.1097/AOG.0b013e3181ab6fd3. PMID 19546755
- [Background] Esteves JS, de Sa RA, de Carvalho PR, Coca Velarde LG. Neonatal outcome in women with preterm premature rupture of membranes (PPROM) between 18 and 26 weeks. J Matern Fetal Neonatal Med. 2016;29(7):1108-12. doi: 10.3109/14767058.2015.1035643. Epub 2015 Jul 3. PMID 26138545
- [Background] Linehan LA, Walsh J, Morris A, Kenny L, O'Donoghue K, Dempsey E, Russell N. Neonatal and maternal outcomes following midtrimester preterm premature rupture of the membranes: a retrospective cohort study. BMC Pregnancy Childbirth. 2016 Jan 29;16:25. doi: 10.1186/s12884-016-0813-3. PMID 26831896
- [Background] Deutsch A, Deutsch E, Totten C, Downes K, Haubner L, Belogolovkin V. Maternal and neonatal outcomes based on the gestational age of midtrimester preterm premature rupture of membranes. J Matern Fetal Neonatal Med. 2010 Dec;23(12):1429-34. doi: 10.3109/14767051003678069. Epub 2010 Mar 17. PMID 20233131
- [Background] Moore T, Hennessy EM, Myles J, Johnson SJ, Draper ES, Costeloe KL, Marlow N. Neurological and developmental outcome in extremely preterm children born in England in 1995 and 2006: the EPICure studies. BMJ. 2012 Dec 4;345:e7961. doi: 10.1136/bmj.e7961. PMID 23212880
- [Background] Kenyon S, Boulvain M, Neilson JP. Antibiotics for preterm rupture of membranes. Cochrane Database Syst Rev. 2013 Dec 2;2013(12):CD001058. doi: 10.1002/14651858.CD001058.pub3. PMID 24297389
- [Background] Mercer BM, Arheart KL. Antimicrobial therapy in expectant management of preterm premature rupture of the membranes. Lancet. 1995 Nov 11;346(8985):1271-9. doi: 10.1016/s0140-6736(95)91868-x. PMID 7475723
- [Background] Kenyon SL, Taylor DJ, Tarnow-Mordi W; ORACLE Collaborative Group. Broad-spectrum antibiotics for preterm, prelabour rupture of fetal membranes: the ORACLE I randomised trial. ORACLE Collaborative Group. Lancet. 2001 Mar 31;357(9261):979-88. doi: 10.1016/s0140-6736(00)04233-1. PMID 11293640
- [Background] Mercer BM, Moretti ML, Prevost RR, Sibai BM. Erythromycin therapy in preterm premature rupture of the membranes: a prospective, randomized trial of 220 patients. Am J Obstet Gynecol. 1992 Mar;166(3):794-802. doi: 10.1016/0002-9378(92)91336-9. PMID 1550145
- [Background] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 statement: updated guidelines for reporting parallel group randomized trials. Ann Intern Med. 2010 Jun 1;152(11):726-32. doi: 10.7326/0003-4819-152-11-201006010-00232. Epub 2010 Mar 24. PMID 20335313
- [Background] Navathe R, Schoen CN, Heidari P, Bachilova S, Ward A, Tepper J, Visintainer P, Hoffman MK, Smith S, Berghella V, Roman A. Azithromycin vs erythromycin for the management of preterm premature rupture of membranes. Am J Obstet Gynecol. 2019 Aug;221(2):144.e1-144.e8. doi: 10.1016/j.ajog.2019.03.009. Epub 2019 Mar 20. PMID 30904320
- [Background] Doyle LW, Crowther CA, Middleton P, Marret S, Rouse D. Magnesium sulphate for women at risk of preterm birth for neuroprotection of the fetus. Cochrane Database Syst Rev. 2009 Jan 21;(1):CD004661. doi: 10.1002/14651858.CD004661.pub3. PMID 19160238
- [Background] DiGiulio DB, Romero R, Kusanovic JP, Gomez R, Kim CJ, Seok KS, Gotsch F, Mazaki-Tovi S, Vaisbuch E, Sanders K, Bik EM, Chaiworapongsa T, Oyarzun E, Relman DA. Prevalence and diversity of microbes in the amniotic fluid, the fetal inflammatory response, and pregnancy outcome in women with preterm pre-labor rupture of membranes. Am J Reprod Immunol. 2010 Jul 1;64(1):38-57. doi: 10.1111/j.1600-0897.2010.00830.x. Epub 2010 Mar 21. PMID 20331587
- [Background] Broekhuizen FF, Gilman M, Hamilton PR. Amniocentesis for gram stain and culture in preterm premature rupture of the membranes. Obstet Gynecol. 1985 Sep;66(3):316-21. PMID 2410839
- [Background] Cotton DB, Hill LM, Strassner HT, Platt LD, Ledger WJ. Use of amniocentesis in preterm gestation with ruptured membranes. Obstet Gynecol. 1984 Jan;63(1):38-43. PMID 6691016
- [Background] Zlatnik FJ, Cruikshank DP, Petzold CR, Galask RP. Amniocentesis in the identification of inapparent infection in preterm patients with premature rupture of the membranes. J Reprod Med. 1984 Sep;29(9):656-60. PMID 6492031
- [Background] Oh KJ, Lee KA, Sohn YK, Park CW, Hong JS, Romero R, Yoon BH. Intraamniotic infection with genital mycoplasmas exhibits a more intense inflammatory response than intraamniotic infection with other microorganisms in patients with preterm premature rupture of membranes. Am J Obstet Gynecol. 2010 Sep;203(3):211.e1-8. doi: 10.1016/j.ajog.2010.03.035. Epub 2010 Aug 3. PMID 20678747
- [Background] Romero R, Emamian M, Quintero R, Wan M, Hobbins JC, Mazor M, Edberg S. The value and limitations of the Gram stain examination in the diagnosis of intraamniotic infection. Am J Obstet Gynecol. 1988 Jul;159(1):114-9. doi: 10.1016/0002-9378(88)90503-0. PMID 2456013
- [Background] Heikkinen T, Laine K, Neuvonen PJ, Ekblad U. The transplacental transfer of the macrolide antibiotics erythromycin, roxithromycin and azithromycin. BJOG. 2000 Jun;107(6):770-5. doi: 10.1111/j.1471-0528.2000.tb13339.x. PMID 10847234
- [Background] Amsden GW. Erythromycin, clarithromycin, and azithromycin: are the differences real? Clin Ther. 1996 Jan-Feb;18(1):56-72; discussion 55. doi: 10.1016/s0149-2918(96)80179-2. PMID 8851453
- [Background] Martinez MA, Vuppalanchi R, Fontana RJ, Stolz A, Kleiner DE, Hayashi PH, Gu J, Hoofnagle JH, Chalasani N. Clinical and histologic features of azithromycin-induced liver injury. Clin Gastroenterol Hepatol. 2015 Feb;13(2):369-376.e3. doi: 10.1016/j.cgh.2014.07.054. Epub 2014 Aug 9. PMID 25111234
- [Background] Russo V, Puzio G, Siniscalchi N. Azithromycin-induced QT prolongation in elderly patient. Acta Biomed. 2006 Apr;77(1):30-2. PMID 16856707
- [Background] Kezerashvili A, Khattak H, Barsky A, Nazari R, Fisher JD. Azithromycin as a cause of QT-interval prolongation and torsade de pointes in the absence of other known precipitating factors. J Interv Card Electrophysiol. 2007 Apr;18(3):243-6. doi: 10.1007/s10840-007-9124-y. Epub 2007 Jun 2. PMID 17546486
- [Background] Ailes EC, Gilboa SM, Gill SK, Broussard CS, Crider KS, Berry RJ, Carter TC, Hobbs CA, Interrante JD, Reefhuis J; and The National Birth Defects Prevention Study. Association between antibiotic use among pregnant women with urinary tract infections in the first trimester and birth defects, National Birth Defects Prevention Study 1997 to 2011. Birth Defects Res A Clin Mol Teratol. 2016 Nov;106(11):940-949. doi: 10.1002/bdra.23570. PMID 27891788
- [Background] Andes D, Craig WA. In vivo activities of amoxicillin and amoxicillin-clavulanate against Streptococcus pneumoniae: application to breakpoint determinations. Antimicrob Agents Chemother. 1998 Sep;42(9):2375-9. doi: 10.1128/AAC.42.9.2375. PMID 9736566
- [Background] Andrew MA, Easterling TR, Carr DB, Shen D, Buchanan ML, Rutherford T, Bennett R, Vicini P, Hebert MF. Amoxicillin pharmacokinetics in pregnant women: modeling and simulations of dosage strategies. Clin Pharmacol Ther. 2007 Apr;81(4):547-56. doi: 10.1038/sj.clpt.6100126. Epub 2007 Feb 28. PMID 17329990
- [Background] Bookstaver PB, Bland CM, Griffin B, Stover KR, Eiland LS, McLaughlin M. A Review of Antibiotic Use in Pregnancy. Pharmacotherapy. 2015 Nov;35(11):1052-62. doi: 10.1002/phar.1649. PMID 26598097
- [Background] Crider KS, Cleves MA, Reefhuis J, Berry RJ, Hobbs CA, Hu DJ. Antibacterial medication use during pregnancy and risk of birth defects: National Birth Defects Prevention Study. Arch Pediatr Adolesc Med. 2009 Nov;163(11):978-85. doi: 10.1001/archpediatrics.2009.188. PMID 19884587
- [Background] Jacobson GF, Autry AM, Kirby RS, Liverman EM, Motley RU. A randomized controlled trial comparing amoxicillin and azithromycin for the treatment of Chlamydia trachomatis in pregnancy. Am J Obstet Gynecol. 2001 Jun;184(7):1352-4; discussion 1354-6. doi: 10.1067/mob.2001.115050. PMID 11408852
- [Background] Lamont HF, Blogg HJ, Lamont RF. Safety of antimicrobial treatment during pregnancy: a current review of resistance, immunomodulation and teratogenicity. Expert Opin Drug Saf. 2014 Dec;13(12):1569-81. doi: 10.1517/14740338.2014.939580. Epub 2014 Sep 5. PMID 25189188
- [Background] Muanda FT, Sheehy O, Berard A. Use of antibiotics during pregnancy and the risk of major congenital malformations: a population based cohort study. Br J Clin Pharmacol. 2017 Nov;83(11):2557-2571. doi: 10.1111/bcp.13364. Epub 2017 Aug 11. PMID 28722171
- [Background] Muller AE, Oostvogel PM, DeJongh J, Mouton JW, Steegers EA, Dorr PJ, Danhof M, Voskuyl RA. Pharmacokinetics of amoxicillin in maternal, umbilical cord, and neonatal sera. Antimicrob Agents Chemother. 2009 Apr;53(4):1574-80. doi: 10.1128/AAC.00119-08. Epub 2009 Jan 21. PMID 19164154
- [Background] Piotin A, Godet J, Trubiano JA, Grandbastien M, Guenard-Bilbault L, de Blay F, Metz-Favre C. Predictive factors of amoxicillin immediate hypersensitivity and validation of PEN-FAST clinical decision rule. Ann Allergy Asthma Immunol. 2022 Jan;128(1):27-32. doi: 10.1016/j.anai.2021.07.005. Epub 2021 Jul 13. PMID 34271183
- [Background] Koosakulchai V, Sangsupawanich P, Wantanaset D, Jessadapakorn W, Jongvilaikasem P, Yuenyongviwat A. Safety of direct oral provocation testing using the Amoxicillin-2-step-challenge in children with history of non-immediate reactions to amoxicillin. World Allergy Organ J. 2021 Jul 9;14(7):100560. doi: 10.1016/j.waojou.2021.100560. eCollection 2021 Jul. PMID 34306301
- [Background] Schrufer P, Brockow K, Stoevesandt J, Trautmann A. Predominant patterns of beta-lactam hypersensitivity in a single German Allergy Center: exanthem induced by aminopenicillins, anaphylaxis by cephalosporins. Allergy Asthma Clin Immunol. 2020 Nov 17;16(1):102. doi: 10.1186/s13223-020-00488-0. PMID 33292467
- [Background] Rodriguez-Martin S, Martin-Merino E, Lerma V, Rodriguez-Miguel A, Gonzalez O, Gonzalez-Herrada C, Ramirez E, Bellon T, de Abajo FJ. Active surveillance of severe cutaneous adverse reactions: A case-population approach using a registry and a health care database. Pharmacoepidemiol Drug Saf. 2018 Sep;27(9):1042-1050. doi: 10.1002/pds.4622. Epub 2018 Jul 27. PMID 30051945
- [Background] Yang MS, Lee JY, Kim J, Kim GW, Kim BK, Kim JY, Park HW, Cho SH, Min KU, Kang HR. Searching for the Culprit Drugs for Stevens-Johnson Syndrome and Toxic Epidermal Necrolysis from a Nationwide Claim Database in Korea. J Allergy Clin Immunol Pract. 2020 Feb;8(2):690-695.e2. doi: 10.1016/j.jaip.2019.09.032. Epub 2019 Oct 12. PMID 31614216
- [Background] Kuehn J, Ismael Z, Long PF, Barker CI, Sharland M. Reported rates of diarrhea following oral penicillin therapy in pediatric clinical trials. J Pediatr Pharmacol Ther. 2015 Mar-Apr;20(2):90-104. doi: 10.5863/1551-6776-20.2.90. PMID 25964726
- [Background] McFarland LV, Ozen M, Dinleyici EC, Goh S. Comparison of pediatric and adult antibiotic-associated diarrhea and Clostridium difficile infections. World J Gastroenterol. 2016 Mar 21;22(11):3078-104. doi: 10.3748/wjg.v22.i11.3078. PMID 27003987
- [Background] Nasiri MJ, Goudarzi M, Hajikhani B, Ghazi M, Goudarzi H, Pouriran R. Clostridioides (Clostridium) difficile infection in hospitalized patients with antibiotic-associated diarrhea: A systematic review and meta-analysis. Anaerobe. 2018 Apr;50:32-37. doi: 10.1016/j.anaerobe.2018.01.011. Epub 2018 Jan 31. PMID 29408016
- [Background] Peled N, Pitlik S, Samra Z, Kazakov A, Bloch Y, Bishara J. Predicting Clostridium difficile toxin in hospitalized patients with antibiotic-associated diarrhea. Infect Control Hosp Epidemiol. 2007 Apr;28(4):377-81. doi: 10.1086/513723. Epub 2007 Mar 9. PMID 17385141
- [Background] Nimrod C, Varela-Gittings F, Machin G, Campbell D, Wesenberg R. The effect of very prolonged membrane rupture on fetal development. Am J Obstet Gynecol. 1984 Mar 1;148(5):540-3. doi: 10.1016/0002-9378(84)90743-9. PMID 6702914
- [Background] Christianson C, Huff D, McPherson E. Limb deformations in oligohydramnios sequence: effects of gestational age and duration of oligohydramnios. Am J Med Genet. 1999 Oct 29;86(5):430-3. PMID 10508984
- [Background] Winn HN, Chen M, Amon E, Leet TL, Shumway JB, Mostello D. Neonatal pulmonary hypoplasia and perinatal mortality in patients with midtrimester rupture of amniotic membranes--a critical analysis. Am J Obstet Gynecol. 2000 Jun;182(6):1638-44. doi: 10.1067/mob.2000.107435. PMID 10871491